CLINICAL TRIAL: NCT03454867
Title: Hemofiltration in Acute Ischemic Stroke Management
Brief Title: Hemofiltration in Acute Ischemic Stroke
Acronym: HAISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Dmitriy Viderman, Attending anesthesiologist & intensivist, University Medical Center, Kazakhstan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemoinstroke
Record Dates: First submitted 2018-02-16; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Hemofiltration

STUDY DESIGN:
Intervention Model Description: Hemofiltration protocol. Hemofiltration was started after all enrollment criteria (informed consent, inclusion/exclusion criteria checklists, registration and assignment to treatment arm) had been met . Vascular access was secured by inserting an 11F double lumen catheter (GamCath, Gambro, Germany) into the jugular, femoral or subclavian vein. CVVH (continuous veno-venous hemofiltration) was carried out using a hemofiltration machine (Fresenius Multifiltrate, Germany). In all patients a 1.9 m2 highly permeable cellulose triacetate hemofilter was used (NIPRO UF205, Nissho corporation, Japan). All patients were treated by CVVH with the predilution mode; the blood flow was set at 180 ml/min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemofiltration (treatment) (Experimental): Standard acute ischemic stroke treatment + hemofiltration Standard treatment included thrombolytic therapy for eligible candidates (tPA 0,9 mg/kg, max dose 90 mg)
  Interventions: Device: Hemofiltration; Procedure: Standard acute ischemic stroke treatment
- Control (Active Comparator): Standard acute ischemic stroke treatment Standard treatment included thrombolytic therapy for eligible candidates (tPA 0,9 mg/kg, max dose 90 mg)
  Interventions: Procedure: Standard acute ischemic stroke treatment

INTERVENTIONS:
Device: Hemofiltration
  Arms: Hemofiltration (treatment)
Procedure: Standard acute ischemic stroke treatment

SUMMARY:
Ischemic stroke is accompanied by a three to four hundred percent increase in the brain's extracellular fluid (ECF) and cerebrospinal fluid (CSF) concentration of glutamate, which diffuses and damages surrounding neurons. In this study we tested our hypothesis that blood glutamate levels can be reduced by hemofiltration, resulting in increased extracellular clearance of glutamate and attenuated neurodegeneration, and that decreased blood glutamate levels can provide significant neuroprotection against stroke-associated neurodegeneration, dysfunction and death. Our primary outcome of interest was to assess safety of hemofiltration in acute ischemic stroke patients.

DETAILED DESCRIPTION:
Ethical Conduct of the Study

Investigator Responsibilities

The principle investigator was responsible for monitoring and responding to adverse events, ethical participant use, compliance with the protocols and any protocol amendments, decisions to end the study early and compliance with data and sample management protocols. CO-PI was trained in both local and international requirements and standards and assisted and report to the PI on these tasks.

Participant Selection and Enrollment

Eligible participants were identified by medical staff at the ICU or emergency department. Enrollment will be standardized and directed by Co-PI.

Screening for Eligibility

A screening log was completed for all eligible patients. Data including inclusion criteria met, exclusion criteria not met and date consent obtained was collected on this form. It was kept in a locked cabinet at the center.

Informed Consent

The informed consent form was available in both Russian and Kazakh languages and was approved by the Institutional Research Ethics Committee (IREC) before use.

Monitoring for safety (hemofiltration-related adverse events (HRAE). All adverse events which occurred during the course of HF including the serious adverse events (SAE) were documented and analyzed. The attending physicians as well as the chief of neurocritical care unit and the principal investigator were responsible for screening for HRAE. In case if any of HRAE occurred all research team members as well as the chief of ICU and the medical director of the hospital were informed. All HRAEs were analyzed by the research team members and the medical director of the hospital. The patients were screened for the following adverse events: hypotension, hypertension, cardiac dysrhythmia, hypothermia or hyperthermia, disorders of water-electrolyte and acid-base balance, bleeding disorders, hemorrhagic transformation of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 year-old; both males and females;
2. Diagnosis of acute ischemic stroke verified by CT or MRI and moderate to severe disability (NIHSS 5-21 points, GCS > 4 points and < 12);
3. Able to start hemofiltration treatment within 12 hours of stroke onset.;
4. Signed written informed consent in either Kazakh or Russian.

Exclusion Criteria:

1. Age below 18 years or above 75 years;
2. Presentation over 12 hours from stroke onset;
3. Decompensated coronary heart disease (unstable angina, acute myocardial infarction, heart failure - according to New York or Canadian classification, 3, blood disorders, known coagulopathy, platelet count less than75 000 / mmc;
4. Pulmonary edema, shock, hemodynamic instability;
5. Intracranial hemorrhage or lesions (brain abscess, tumors);
6. Inability to obtain informed consent;
7. Pregnancy;
8. Contraindications for CT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Safety monitoring for adverse events | 28 days
  The patients were screened continuously for the following adverse events: death, bleeding disorders, hemorrhagic transformation of acute ischemic stroke, central line-related blood stream infection, cardiac dysrhythmia within 28 days

IPD SHARING:
Plan to Share IPD: No
We will work on method of data sharing